CLINICAL TRIAL: NCT02545543
Title: A Phase 3, Randomized, Multicenter, Observer-Blinded, Noninferiority Study to Evaluate the Immunogenicity and Safety of a Seqirus Quadrivalent Inactivated Influenza Virus Vaccine (Seqirus QIV) With a US-Licensed 2015-2016 Quadrivalent Inactivated Comparator Influenza Vaccine (Comparator QIV) in a Pediatric Population 5 Through 17 Years of Age
Brief Title: A Study to Evaluate the Immunogenicity and Safety of Seqirus Quadrivalent Influenza Vaccine (QIV) in a Pediatric Population 5 Through 17 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSLCT-QIV-13-02
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Seqirus Quadrivalent Inactivated Influenza Vaccine (Experimental): The Seqirus study vaccine is a sterile, thimerosal-free suspension containing 60 mcg total hemagglutinin antigen per 0.5 mL dose (15 mcg each of the four recommended influenza strains for the Northern Hemisphere 2015/2016 influenza season).
  Interventions: Biological: Seqirus QIV
- Comparator Quadrivalent Influenza Vaccine (Active Comparator): The comparator Quadrivalent Inactivated Influenza vaccine is a US-licensed product containing four recommended influenza strains for the Northern Hemisphere 2015/2016 influenza season.
  Interventions: Biological: Comparator QIV

INTERVENTIONS:
Biological: Seqirus QIV — Seqirus QIV, inactivated, split-virion, thimerosal-free, quadrivalent influenza vaccine, administered as a 0.5 mL intramuscular dose. The vaccine is presented in a prefilled needleless syringe.
  The subject's age and influenza vaccination history determines the dosing regimen (a single vaccination or a 2-vaccination regimen administered 28 days apart) according to the most recent US ACIP guidelines for seasonal influenza vaccination.
  Arms: Seqirus Quadrivalent Inactivated Influenza Vaccine
Biological: Comparator QIV — The US-licensed Comparator QIV, inactivated, split-virion, thimerosal-free, quadrivalent influenza vaccine, administered as a 0.5 mL intramuscular dose. The vaccine is presented in a prefilled needleless syringe.
  The subject's age and influenza vaccination history determines the dosing regimen (a single vaccination or a 2-vaccination regimen administered 28 days apart) according to the most recent US ACIP guidelines for seasonal influenza vaccination.
  Other Names: Fluarix Quadrivalent
  Arms: Comparator Quadrivalent Influenza Vaccine

SUMMARY:
This is a study to assess the immune (antibody) response and safety of a Seqirus split virion, inactivated Quadrivalent Influenza Vaccine (Seqirus QIV), in comparison with a US licensed 2015/2016 Quadrivalent Influenza Vaccine (comparator QIV) in a healthy pediatric population 5 through 17 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 5 through 17 years of age on the day of first study vaccination.
* Parent or legally acceptable representative able to provide written informed consent and be willing and able to adhere to all protocol requirements including blood draws. Participant assent will also be obtained if required.
* If applicable, females of childbearing potential (ie, ovulating, not surgically sterile) must be abstinent or be willing to use a medically accepted contraceptive regimen until at least 28 days after the last Study Vaccine. Females of childbearing potential must return a negative urine pregnancy test result, prior to any vaccination dose with the Study Vaccine.

Exclusion Criteria:

* History of allergic reactions to egg proteins or any components of the Study Vaccines.
* History of serious adverse reactions to any influenza vaccines.
* History of Guillain-Barré syndrome or other demyelinating disease.
* History of licensed or investigational influenza vaccination in the last 6 months.
* Clinical signs of active infection and/or an oral temperature of ≥ 100°F (37.8°C) on the day of planned Study Vaccine administration or within 48 hours preceding vaccination.
* Current or recent, acute or chronic medical conditions that in the opinion of the Investigator are clinically significant and/or unstable (such as illness exacerbations) within the preceding 30 days.
* History of any seizures, with the exception of a single febrile seizure.
* Self-reported or known seropositivity suggestive of acute or chronic viral infection for human immunodeficiency virus, hepatitis B or hepatitis C.
* Known or suspected congenital or acquired immunosuppressive conditions.
* Current or recent immunosuppressive or immunomodulatory therapy, as follows:

  * Chronic or long-term systemic corticosteroids: ≥ 0.125 mg/kg/day of oral prednisolone or equivalent daily;
  * Sporadic systemic corticosteroids: ≥ 0.5 mg/kg/day of oral prednisolone or equivalent for two or more short courses of > 3 days in the 3 months preceding vaccination;
  * Antineoplastic chemotherapy or radiation therapy within the 6 months preceding vaccination.

Note: Use of topical, inhalant or localised tissue injections of corticosteroids prior to administration of the Study Vaccine or throughout the study are acceptable.

* Administration of immunoglobulin and/or any blood products within the 3 months preceding vaccination, or planned administration during the study.
* Participation in a clinical trial or use of an investigational compound within 28 days prior to the first dose of Study Vaccine, or within 28 days after receiving the final indicated dose of Study Vaccine, or plans to enter a study during this period.
* Vaccination with a licensed vaccine 28 days (for live or inactivated vaccines) prior to receiving the first dose of Study Vaccine, or plans to receive any licensed vaccine prior to the Study Exit Visit.
* Pregnant or lactating females.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2278 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Physician Seqirus, Study Director — Seqirus
Locations (32):
- United States (32):
  - Site 296, Huntsville, Alabama
  - Site 401, Madera, California
  - Site 397, Ontario, California
  - Site 392, Redding, California
  - Site 402, Sacramento, California
  - Site 398, San Jose, California
  - Site 388, Hialeah, Florida
  - Site 293, Melbourne, Florida
  - Site 289, Boise, Idaho
  - Site 294, Peoria, Illinois
  - Site 390, Augusta, Kansas
  - Site 396, Newton, Kansas
  - Site 400, Park City, Kansas
  - Site 317, Wichita, Kansas
  - Site 386, Bardstown, Kentucky
  - Site 393, Metairie, Louisiana
  - Site 287, St Louis, Missouri
  - Site 316, Bellevue, Nebraska
  - Site 382, Omaha, Nebraska
  - Site 285, Binghamton, New York
  - Site 387, Cary, North Carolina
  - Site 385, Cincinnati, Ohio
  - Site 383, Cleveland, Ohio
  - Site 399, Dayton, Ohio
  - Site 384, Grove City, Ohio
  - Site 389, Gresham, Oregon
  - Site 283, Austin, Texas
  - Site 282, Fort Worth, Texas
  - Site 288, San Angelo, Texas
  - Site 394, San Antonio, Texas
  - Site 395, Layton, Utah
  - Site 300, Salt Lake City, Utah

REFERENCES:
- [Derived] Airey J, Albano FR, Sawlwin DC, Jones AG, Formica N, Matassa V, Leong J. Immunogenicity and safety of a quadrivalent inactivated influenza virus vaccine compared with a comparator quadrivalent inactivated influenza vaccine in a pediatric population: A phase 3, randomized noninferiority study. Vaccine. 2017 May 9;35(20):2745-2752. doi: 10.1016/j.vaccine.2017.03.028. Epub 2017 Apr 5. PMID 28390934

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 14-SEP-2015, Last Patient Last Visit: 13-JUN-2016. Number of activated sites that enrolled subjects: 32 (all based in USA).
Pre-assignment Details: Number of subjects screened: 2349. Number of subjects randomized: 2278
Groups:
- Seqirus Quadrivalent Influenza Vaccine: The Seqirus study vaccine is a sterile, thimerosal-free suspension containing 60 mcg total hemagglutinin antigen per 0.5 mL dose (15 mcg each of the four recommended influenza strains for the Northern Hemisphere 2015/2016 influenza season).
  Seqirus QIV: Seqirus QIV, inactivated, split-virion, thimerosal-free, quadrivalent influenza vaccine, administered as a 0.5 mL intramuscular dose. The vaccine is presented in a prefilled needleless syringe.
  The subject's age and influenza vaccination history determines the dosing regimen (a single vaccination or a 2-vaccination regimen administered 28 days apart) according to the most recent US ACIP guidelines for seasonal influenza vaccination.
- Comparator Quadrivalent Influenza Vaccine: The comparator Quadrivalent Inactivated Influenza vaccine is a US-licensed product containing four recommended influenza strains for the Northern Hemisphere 2015/2016 influenza season.
  Comparator QIV: The US-licensed Comparator QIV, inactivated, split-virion, thimerosal-free, quadrivalent influenza vaccine, administered as a 0.5 mL intramuscular dose. The vaccine is presented in a prefilled needleless syringe.
  The subject's age and influenza vaccination history determines the dosing regimen (a single vaccination or a 2-vaccination regimen administered 28 days apart) according to the most recent US ACIP guidelines for seasonal influenza vaccination.
Period: Overall Study
Arm/Group | Seqirus Quadrivalent Influenza Vaccine | Comparator Quadrivalent Influenza Vaccine
Started | 1709 | 569
Completed | 1628 | 535
Not Completed | 81 | 34
Not completed — Lost to Follow-up | 67 | 25
Not completed — Physician Decision | 3 | 0
Not completed — Withdrawal by Subject | 9 | 8
Not completed — Noncomplaince | 1 | 0
Not completed — Enrolment of subject at >1 study site | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) was used for analysis of subject characteristics and comprised all subjects who gave informed consent and who were randomized to treatment. Screening failures were not included in the FAS.
Groups:
- Total: Total of all reporting groups
Arm/Group | Seqirus Quadrivalent Influenza Vaccine | Comparator Quadrivalent Influenza Vaccine | Total
Number analyzed (Participants) | 1709 | 569 | 2278
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.5 (3.49) | 9.5 (3.46) | 9.5 (3.48)
Age, Customized [Count of Participants; unit: Participants]
  5 through 8 years | 875 | 291 | 1166
  9 through 17 years | 834 | 278 | 1112
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 825 | 267 | 1092
  Male | 884 | 302 | 1186
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 412 | 130 | 542
  Not Hispanic or Latino | 1293 | 438 | 1731
  Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 2 | 7
  Asian | 16 | 2 | 18
  Native Hawaiian or Other Pacific Islander | 13 | 2 | 15
  Black or African American | 359 | 113 | 472
  White | 1239 | 430 | 1669
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 77 | 20 | 97
Region of Enrollment [Number; unit: participants]
  United States | 1709 | 569 | 2278

OUTCOME MEASURES:

1. Primary Outcome: The Geometric Mean Titer (GMT) Ratio of Each Virus Strain.
Description: Noninferiority of Seqirus QIV compared to comparator QIV was assessed by the eight co-primary endpoints of hemagglutination inhibition (HI) antibody geometric mean titer (GMT) and seroconversion rate (SCR) for each viral strain included in the vaccines. The GMT ratio is defined as the geometric mean of the postvaccination HI titer for the US-licensed comparator QIV over the geometric mean of the postvaccination HI titer for Seqirus QIV.
Time Frame: 28 days after last vaccination.
Population: The Per Protocol Population was used for the primary and secondary analysis of immunogenicity data and included subjects in the Evaluable Population minus any subjects with deviations that were thought to potentially affect the immunogenicity results, following medical review prior to unblinding.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- GMT Ratios: GMT Comparator QIV Over GMT Seqirus QIV: GMT Ratios: GMT Comparator Quadrivalent Influenza Vaccine over GMT Seqirus Quadrivalent Influenza Vaccine
Arm/Group | GMT Ratios: GMT Comparator QIV Over GMT Seqirus QIV
Number analyzed (Participants) | 2133
Ratio
  A/H1N1 | 1.01 [0.93 to 1.09]
  A/H3N2 | 1.05 [0.96 to 1.15]
  B/Yamagata | 0.89 [0.81 to 0.98]
  B/Victoria | 0.92 [0.83 to 1.02]

2. Primary Outcome: The Difference in Seroconversion Rate (SCR) for Each Virus Strain.
Description: Noninferiority of Seqirus QIV compared to Comparator QIV was assessed by the eight co-primary endpoints of HI geometric mean titer (GMT) and seroconversion rate (SCR) for each viral strain. The rate of SCR is defined as the percentage of subjects with either a prevaccination HI titer < 1:10 and a postvaccination HI titer ≥ 1:40, or a prevaccination HI titer ≥ 1:10 and a ≥ 4-fold increase in postvaccination HI titer. For the SCR comparison, the difference between the SCR for each virus strain will be determined.
Time Frame: 28 days after last vaccination.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SCR Difference = Comparator QIV SCR % Minus Seqirus QIV SCR %: Seroconversion rate difference = Comparator QIV SCR percentage minus Seqirus QIV SCR percentage
Arm/Group | SCR Difference = Comparator QIV SCR % Minus Seqirus QIV SCR %
Number analyzed (Participants) | 2133
percentage of participants
  A/H1N1 | -3.1 [-8.0 to 1.8]
  A/H3N2 | 0.4 [-4.5 to 5.3]
  B/Yamagata | -3.4 [-8.3 to 1.5]
  B/Victoria | -2.0 [-6.9 to 2.9]

3. Secondary Outcome: Safety Endpoint: The Frequency and Severity of Solicited Local Adverse Reactions.
Description: Frequency and severity of solicited local adverse reactions (AEs) for 7 days (ie, day of vaccination and 6 subsequent days) after each vaccination dose
Time Frame: 7 days after each vaccination.
Population: The Solicited Safety Population comprises all subjects in the FAS who received at least one dose or partial dose of Study Vaccine and provided any evaluable data on solicited events.
Measure: Number; unit: participants
Arm/Group | Seqirus Quadrivalent Influenza Vaccine | Comparator Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 1621 | 535
participants
  Frequency of Solicited Local AEs | 909 | 279
  Severe (Grade 3) Solicited Local AEs | 71 | 21

4. Secondary Outcome: Safety Endpoint: The Frequency and Severity of Solicited Systemic Adverse Events (AEs).
Description: Frequency and severity of solicited systemic adverse events (AEs) for 7 days (ie, day of vaccination and 6 subsequent days) after each vaccination dose
Time Frame: 7 days after each vaccination.
Population: The Solicited Safety Population comprised all subjects in the FAS who received at least one dose or partial dose of Study Vaccine and provided any evaluable data on solicited events.
Measure: Number; unit: participants
Arm/Group | Seqirus Quadrivalent Influenza Vaccine | Comparator Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 1621 | 535
participants
  Frequency of Solicited Systemic AEs | 499 | 147
  Severe (Grade 3) Solicited Systemic AEs | 24 | 6

5. Secondary Outcome: Safety Endpoint: The Frequency of Cellulitis-like Reaction.
Description: Frequency of cellulitis-like reaction for at least 28 days after each vaccination dose
Time Frame: 28 days after each vaccination.
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Seqirus Quadrivalent Influenza Vaccine | Comparator Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 1621 | 535
participants | 1 | 0

6. Secondary Outcome: Safety Endpoint: The Frequency and Severity of Unsolicited Adverse Events (AEs).
Description: Frequency and severity of unsolicited AEs for at least 28 days (ie, day of vaccination and 27 subsequent days) after each vaccination dose
Time Frame: 28 days after each vaccination.
Population: The Overall Safety Population comprises all subjects in the FAS who received at least one dose or partial dose of Study Vaccine and provided any evaluable follow-up safety data.
Measure: Number; unit: participants
Arm/Group | Seqirus Quadrivalent Influenza Vaccine | Comparator Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 1692 | 560
participants
  At least one Unsolicited AE | 269 | 70
  Severe (Grade 3) Unsolicited AE | 11 | 6

7. Secondary Outcome: Safety Endpoint: The Frequency of Serious Adverse Events (SAEs).
Description: Frequency of serious adverse events (SAEs) for 180 days after the last vaccination dose.
Time Frame: 180 days after the last vaccination dose.
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Seqirus Quadrivalent Influenza Vaccine | Comparator Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 1692 | 560
participants | 8 | 2

8. Secondary Outcome: Immunogenicity Endpoint: GMTs - Geometric Mean of HI Titers Prevaccination (Day 1) and Postvaccination (Study Exit Visit)
Description: The humoral immune response was assessed for Seqirus QIV & comparator QIV. Serum HI titers against the 4 influenza vaccine strains was used to calculate:
  - Geometric mean of HI titers prevaccination & postvaccination
Time Frame: 28 days after last vaccination.
Population: The Per-Protocol Population comprised all subjects in the Evaluable Population who did not have any protocol deviations that were medically assessed as potentially impacting on immunogenicity results
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Seqirus Quadrivalent Influenza Vaccine | Comparator Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 1605 | 528
Titer
  A/H1N1 (pre-vaccination) | 114.8 [106.79 to 123.33] | 119.5 [105.48 to 135.38]
  A/H3N2 (pre-vaccination) | 75.2 [70.80 to 79.88] | 72.1 [64.61 to 80.40]
  B/Yamagata (pre-vaccination) | 10.5 [10.12 to 10.99] | 10.4 [9.69 to 11.22]
  B/Victoria (pre-vaccination) | 17.0 [16.10 to 17.85] | 16.9 [15.42 to 18.46]
  A/H1N1 (post-vaccination) | 858.7 [821.46 to 897.65] | 875.1 [814.14 to 940.59]
  A/H3N2 (post-vaccination) | 803.6 [763.01 to 846.26] | 825.6 [756.12 to 901.55]
  B/Yamagata (post-vaccination) | 60.7 [57.52 to 64.01] | 54.3 [49.65 to 59.28]
  B/Victoria (post-vaccination) | 140.9 [132.97 to 149.26] | 130.3 [117.07 to 145.06]

9. Secondary Outcome: Immunogenicity Endpoint: Seroconversion Rate (SCR)
Description: The humoral immune response was assessed for Seqirus QIV & comparator QIV. Serum HI titers against the 4 influenza vaccine strains was used to calculate:
  - SCRs: % of subjects with either a prevaccination HI titer < 1:10 and a postvaccination HI titer ≥ 1:40 or a prevaccination titer ≥ 1:10 and a ≥ 4-fold increase in postvaccination titer
Time Frame: 28 days after last vaccination.
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Seqirus Quadrivalent Influenza Vaccine | Comparator Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 1605 | 528
percentage of participants
  A/H1N1 | 66.4 [64.0 to 68.7] | 63.3 [59.0 to 67.4]
  A/H3N2 | 82.9 [81.0 to 84.7] | 83.3 [79.9 to 86.4]
  B/Yamagata | 58.5 [56.0 to 60.9] | 55.1 [50.8 to 59.4]
  B/Victoria | 72.1 [69.8 to 74.3] | 70.1 [66.0 to 74.0]

10. Secondary Outcome: Immunogenicity Endpoint: Seroprotection Rate
Description: The humoral immune response was assessed for Seqirus QIV & comparator QIV. Serum HI titers against the 4 influenza vaccine strains was used to calculate:
  - The % of subjects with a titer ≥40 (seroprotection rates) at Day 1 and at Exit Visit
Time Frame: 28 days after last vaccination.
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Seqirus Quadrivalent Influenza Vaccine | Comparator Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 1605 | 528
percentage of participants
  A/H1N1 (pre-vaccination) | 81.2 [79.2 to 83.1] | 82.0 [78.5 to 85.2]
  A/H3N2 (pre-vaccination) | 76.7 [74.6 to 78.7] | 74.2 [70.3 to 77.9]
  B/Yamagata (pre-vaccination) | 13.0 [11.4 to 14.7] | 14.2 [11.3 to 17.5]
  B/Victoria (pre-vaccination) | 27.9 [25.7 to 30.2] | 27.8 [24.1 to 31.9]
  A/H1N1 (post-vaccination) | 99.7 [99.3 to 99.9] | 99.6 [98.6 to 100.0]
  A/H3N2 (post-vaccination) | 99.4 [98.9 to 99.7] | 99.4 [98.3 to 99.9]
  B/Yamagata (post-vaccination) | 75.0 [72.8 to 77.1] | 74.2 [70.3 to 77.9]
  B/Victoria (post-vaccination) | 90.3 [88.7 to 91.7] | 88.6 [85.6 to 91.2]

11. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Fold Increase (GMFI)
Description: The humoral immune response was assessed for Seqirus QIV & comparator QIV. Serum HI titers against the 4 influenza vaccine strains was used to calculate:
  - Geometric mean fold increase (GMFI): geometric mean fold titer rise from Day 1 to Exit Visit
Time Frame: 28 days after last vaccination.
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change Titer (GMFI)
Arm/Group | Seqirus Quadrivalent Influenza Vaccine | Comparator Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 1605 | 528
Fold Change Titer (GMFI)
  A/H1N1 | 7.5 [6.99 to 8.01] | 7.3 [6.46 to 8.30]
  A/H3N2 | 10.7 [10.09 to 11.31] | 11.5 [10.32 to 12.71]
  B/Yamagata | 5.8 [5.44 to 6.08] | 5.2 [4.75 to 5.71]
  B/Victoria | 8.3 [7.81 to 8.84] | 7.7 [6.92 to 8.62]

ADVERSE EVENTS:
Time Frame: Local and systemic solicited AEs collected from Day 1 to Day 7. Unsolicited AEs collected for 28 days after each vaccination dose. SAEs collected for 180 days after last vaccination.
Groups:
- Seqirus Quadrivalent Influenza Vaccine: The Seqirus study vaccine is a sterile, thiomersal-free suspension containing 60 mcg total hemagglutinin antigen per 0.5 mL dose (15 mcg each of the four recommended influenza strains for the Northern Hemisphere 2015/2016 influenza season).
  Seqirus QIV: Seqirus QIV, inactivated, split-virion, thimerosal-free, quadrivalent influenza vaccine, administered as a 0.5 mL intramuscular dose. The vaccine is presented in a prefilled needleless syringe.
  The subject's age and influenza vaccination history determines the dosing regimen (a single vaccination or a 2-vaccination regimen administered 28 days apart) according to the most recent US ACIP guidelines for seasonal influenza vaccination.
Arm/Group | Seqirus Quadrivalent Influenza Vaccine | Comparator Quadrivalent Influenza Vaccine
Serious Adverse Events (participants affected / at risk) | 8/1692 | 2/560
Other Adverse Events (participants affected / at risk) | 1019/1692 | 319/560
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Seqirus Quadrivalent Influenza Vaccine (N=1692) | Comparator Quadrivalent Influenza Vaccine (N=560)
Gasteritis viral (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Pancreatic injury (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Seqirus Quadrivalent Influenza Vaccine (N=1692) | Comparator Quadrivalent Influenza Vaccine (N=560)
Pain (General disorders) | 833 | 254
Swelling (General disorders) | 224 | 62
Redness (General disorders) | 278 | 93
Nausea (Gastrointestinal disorders) | 120 | 44
Diarrhea (Gastrointestinal disorders) | 86 | 21
Headache (Nervous system disorders) | 251 | 67
Myalgia (Musculoskeletal and connective tissue disorders) | 213 | 60
Malasia and Fatigue (General disorders) | 152 | 36
Fever (General disorders) | 54 | 12
Vomiting (Gastrointestinal disorders) | 34 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Seqirus agreements and restrictions on publishing may vary with individual investigators; however, Seqirus will not prohibit any investigator from publishing. Seqirus supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.